CLINICAL TRIAL: NCT03607474
Title: Patient and Partner Perception After Remission of Cushing's Syndrome - Parathyroid 3 Cushing Study
Brief Title: Patient and Partner Perception After Remission of Cushing's Syndrome
Acronym: CUSHING
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-38
Record Dates: First submitted 2018-06-28; First posted 2018-07-31 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Hypercorticism
MeSH Terms: conditions — Adrenocortical Hyperfunction | interventions — Caregivers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Couple (Patients and caregivers): Patient in remission of hypercortisolism Caregivers will be the spouse or, failing that, a person close to the patient, who has been in regular contact with the patient since taking care of him.
  Questionnaires of life quality for patients Questionnaires of life quality for caregivers
  Interventions: Other: Questionnaires of life quality for patients; Other: Questionnaires of life quality for caregivers

INTERVENTIONS:
Other: Questionnaires of life quality for patients — * the WhoQoL
  * a specific scale of Cushing's syndrome
  * The Beck II scale
  * HAD scale
  * Rosenberg questionnaire
  * Stunkard, Sorensen and Schlusinger (1983) figurines
  * Brief Cope scale
Other: Questionnaires of life quality for caregivers — * the WhoQoL
  * The Beck II scale
  * HAD scale

SUMMARY:
Hypercortisolism leads to long term physical and cognitive sequelae. This also holds true for quality of life, even several years after remission. This altered quality of life, highly subjective, is however, badly evaluated by the family of the patient. This could lead to misunderstanding, avec worsen the general physical and mental health of the patient. To our knowledge, this theoretical difference of perception has never been evaluated up to now.

The aim of our study is to evaluate the difference of perception of the quality of life and body image between patients in remission of hypercortisolism, and their caregivers. Secondary objectives will be to evaluate the quality of life of the caregivers, the coping strategies, and the depression/anxiety parameters of both the patient and the caregiver. Patients and methods: the study is Observative, prospective and non-randomized. Inclusion criteria will be patients, aged more than 18, with hypercortisolism in remission for at least 1 year. Self-questionnaires on quality of life, body image, coping, depression and anxiety will be provided to the patient and his/her caregiver. Fulfilling will be blind between the patient and his/her caregiver. Inclusion period will be 12 months.

Results will be compared between the patient and his/her caregiver. Expected results: investigators anticipate that some caregivers will have a different perception of the general physical and mental condition as stated by the patient. The first time that the quality of life of the caregiver would be also altered.

This original project might lead to modify the management of Cushing's syndrome, by considering both the patient and his/her caregiver on a long term basis after remission.

DETAILED DESCRIPTION:
Introduction: Hypercortisolism leads to long term physical and cognitive sequelae. This also holds true for quality of life, even several years after remission. This altered quality of life, highly subjective, is however, badly evaluated by the family of the patient. This could lead to misunderstanding, avec worsen the general physical and mental health of the patient. To our knowledge, this theoretical difference of perception has never been evaluated up to now. Aims: The aim of our study is to evaluate the difference of perception of the quality of life and body image between patients in remission of hypercortisolism, and their caregivers. Secondary objectives will be to evaluate the quality of life of the caregivers, the coping strategies, and the depression/anxiety parameters of both the patient and the caregiver. Patients and methods: the study is Observative, prospective and non-randomized. Inclusion criteria will be patients, aged more than 18, with hypercortisolism in remission for at least 1 year. Self-questionnaires on quality of life, body image, coping, depression and anxiety will be provided to the patient and his/her caregiver. Fulfilling will be blind between the patient and his/her caregiver. Inclusion period will be 12 months. Results will be compared between the patient and his/her caregiver. Expected results: investigators anticipate that some caregivers will have a different perception of the general physical and mental condition as stated by the patient. The first time that the quality of life of the caregiver could be also altered. Perspectives: This original project might lead to modify the management of Cushing's syndrome, by considering both the patient and his/her caregiver on a long term basis after remission.

ELIGIBILITY:
Inclusion Criteria:

* Subject, male or female over 18
* Subject presenting a hypercortisolism in remission or controlled by a drug treatment for more than one year.
* Subject with a good understanding of the French language
* Non-institutionalized subject
* Subject whose informed consent could be obtained

Exclusion Criteria:

* Minor subject or over 80 years
* Subject presenting hypercortisolism in remission for more than 20 years
* Major cognitive impairment that does not allow answering a questionnaire
* Genetic syndrome responsible for hypercortisolism
* Mixed adenoma whose corticotropic share is responsible for hypercortisolism
* Pituitary carcinoma
* Subject refusing to participate in the study
* Subject having no close
* Subject whose relative refuses to answer the questionnaires

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients, aged more than 18, with hypercortisolism in remission for at least 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
assessment of quality of life | 30 minutes
  the World health organisation Quality Of Life ( WHOQOL) is a specific scale of Cushing's syndrome studying: Physical health (Activities of daily living, Dependence on medicinal substances and medical aids, Energy and fatigue, Mobility, Pain and discomfort, Sleep and rest, Work Capacity) Psychological (Bodily image and appearance, Negative feelings, Positive feelings, Self-esteem, Spirituality / Religion / Personal beliefs, Thinking, learning, memory and concentration Social relationships (Personal relationships, Social support, Sexual activity) Environment (Financial resources, Freedom, physical safety and security, Health and social care, Home environment, Opportunities for acquiring new information and skills, Participation in and opportunities for recreation / leisure activities, Physical environment, Transport) intensity of items is rated from not at all (=0), a little (=1), moderately (=2), very much (=3) to extremely (=4).
anxiety | 30 minutes
  using the Hospital Anxiety and Depression scale The HAD scale is an instrument for detecting anxiety and depressive disorders. It has 14 listed items from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), allowing thus obtaining two scores (maximum score of each score = 21)
  0- never
  1. sometimes
  2. Often enough
  3. very often
body image | 30 minutes
  using the Scale of Estime of Self of Rosenberg:
  10 questions for which it must be indicated how true it is (rated from 1 to 4). Then, simply add your scores to questions 1, 2, 4, 6 and 7. For questions 3, 5, 8, 9 and 10, the quotation is reversed, that is to say, it is necessary to count 4 if you surround the number 1, 3 if you surround the 2, 2 if you surround the 3 and 1 if you surround the 4.
  results: If score below 25, self-esteem is very low. Work in this area seems desirable. If score between 25 and 31, self-esteem is low. Work in this area would be beneficial. If score between 31 and 34, self-esteem is average. If score between 34 and 39, your self-esteem is strong. If score above 39, self-esteem is very high and you tend to be strongly affirmed.
depression | 30 minutes
  The Beck Depression Inventory-II (BDI-II):
  21-item self-report multiple-choice inventory (10 minutes to complete) Widely used indicator of the severity of depression 21 items of symptoms and attitudes graduated from 0 to 3 reflecting the severity of the symptom.
  The maximum total score is 63. score indicates 0-13 minimal depression 14-19: mild depression 20-28 moderate depression 29-63 severe depression
coping | 30 minutes
  Stunkard, Sorensen and Schlusinger (1983) figurines that measure the visual representation of the body The Stunkard scale consists of 9 silhouette figures that increase gradually in size from very thin (a value of 1) to very obese (a value of 9) Self body size is the number of the figure selected by participants in response to the prompt: "Choose the figure that reflects how you think you look." Ideal body size is the number of the figure chosen in response to the prompt: "Choose your ideal figure." For self body size and ideal body size, dummy variables were created for the underweight, normal weight, overweight, and obese body size categories.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM DRIC
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France